CLINICAL TRIAL: NCT04872478
Title: An Open Label Evaluation Phase 1 Trial of the Safety and Pharmacokinetics of MRX-2843 in Adolescents and Adults With Relapsed/Refractory Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, or Mixed Phenotype Acute Leukemia
Brief Title: Pharmacokinetic and Safety Study of MRX-2843 in Adolescents and Adults With Relapsed/Refractory AML, ALL, or MPAL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Meryx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2843-1003
Record Dates: First submitted 2021-04-29; First posted 2021-05-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Mixed Phenotype Acute Leukemia
Keywords: MerTK Inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute | interventions — MRX-2843

STUDY DESIGN:
Intervention Model Description: Patients will be accrued using a 3+3 approach. Cohorts will be escalated based on review of safety data for each patient and cohort.
  The highest dose level administered prior to the dose in which ≥ 33% of patients experience a dose-limiting toxicity [DLT]) will be defined as the MTD. Based on PK, pharmacodynamic data, efficacy, safety and patient tolerability, a recommended dose for further development (RP2D) may be identified that is less than the formal MTD. A dose expansion arm of approximately 12 patients (with 6 patients being FLT3 ITD+ and 6 patients being Mer+/FLT3 WT) will be accrued to further evaluate patients at the RP2D.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation - Level 1 (Experimental): MRX-2843 capsules, QD - 28 day cycles
  Interventions: Drug: MRX-2843
- Dose Escalation - Level 2 (Experimental): MRX-2843 capsules, QD - 28 day cycles
  Interventions: Drug: MRX-2843
- Dose Escalation - Level 3 (Experimental): MRX-2843 capsules, QD - 28 day cycles
  Interventions: Drug: MRX-2843
- Dose Escalation - Level 4 (Experimental): MRX-2843 capsules, QD - 28 day cycles
  Interventions: Drug: MRX-2843
- Dose Escalation - Level 5 (Experimental): MRX-2843 capsules, QD - 28 day cycles
  Interventions: Drug: MRX-2843
- Expansion Arm at RP2D (Experimental): MRX-2843 capsules, QD - 28 day cycles
  Interventions: Drug: MRX-2843

INTERVENTIONS:
Drug: MRX-2843 — MRX-2843 capsules

SUMMARY:
This is a Phase I, open-label, non-randomized, dose escalation study in adolescents and adults with relapsed/refractory acute myeloid leukemia, acute lymphoblastic leukemia, or mixed phenotype acute leukemia. Patients will receive continuous oral MRX-2843 in 28 day cycles at predefined dose cohorts.

DETAILED DESCRIPTION:
This is a Phase I, open-label, non-randomized, dose escalation study in up to 50 adolescent or adult patients with relapsed/refractory acute myeloid leukemia, acute lymphoblastic leukemia, or mixed phenotype acute leukemia. Patients will receive a single dose of MRX-2843 followed by continuous oral MRX-2843 in 28 day cycles at predefined dose cohorts.

A dose expansion arm of approximately 12 patients (with 6 patients being FLT3 ITD+ and 6 patients being Mer+/FLT3 WT) will be accrued to further evaluate patients at the RP2D.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or female at least 12 years of age.
* Patient must weigh at least 40 Kg.
* Patient has histologically or cytologically confirmed diagnosis of AML as defined by the World Health Organization (WHO) criteria (2017), ALL, or MPAL and is in second or later relapse or is refractory to at least one induction regimen.
* The effects of MRX-2843 on developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to remain abstinent, or agree to practice double barrier forms of birth control in which 2 of the following precautions are used during the study and for 4 months after last dose of study drug(s): vasectomy, tubal ligation (or other transcervical sterilization procedures), vaginal diaphragm, intrauterine device, birth control pills, birth control implant, or condom or sponge with spermicide.
* Female patients of childbearing potential must be nonpregnant, nonlactating, and have a negative pregnancy test result at Screening and a negative pregnancy test on Day 1 of Cycles 1-4.
* Patient is able to provide written, informed consent or assent for patients < 18 years of age is provided along with parent/guardian consent before initiation of any study related procedures, and patient is able, in the opinion of the investigator, to comply with all the requirements of the study.
* Patient is able to swallow oral medication.
* Patient has white blood cell (WBC) lower than 25,000/mm3 at Screening prior to initiation of MRX-2843. Patients who are otherwise medically eligible for enrollment but have WBC above 25,000/mm3 are allowed concurrent treatment with hydroxyurea to stabilize the WBC. In these situations, hydroxyurea will be discontinued once WBC is below 10,000/mm3 and at least 1 day prior to start of study treatment. Treatment with hydroxyurea will be allowed during Cycle 1 if deemed needed by the Investigator.
* The Patient has laboratory values at Screening:

  1. Bilirubin ≤ 1.5 the upper limit of normal (ULN). For patients with documented Gilbert's disease, bilirubin ≤ 3.0 mg/dL
  2. Creatinine clearance (CrCl) ≥ 60 mL/min. For creatinine clearance estimation, the Cockcroft and Gault equation should be used:

     Male: CrCl (mL/min) = (140 - age) × wt (kg) / (serum creatinine × 72) (For females: Multiply above result by 0.85)
  3. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN
* Patient has Eastern Cooperative Oncology Group (ECOG) performance status 0-2 or Lansky/Karnofsky ≥ 50.
* For the FLT3ITD expansion cohort at RP2D, the FLT3ITD+ patients should have previously been treated with at least one FLT3 inhibitor prior to enrollment.

Exclusion Criteria:

* To be eligible for this study, each of the following criteria must be satisfied with a "NO" answer:

All Subjects:

* Patient has diagnosis of acute promyelocytic leukemia (or AML M3).
* Patients with known active CNS leukemia.
* Patient has any surgical or medical condition (active or chronic) that may interfere with drug absorption, distribution, metabolism, or excretion of the study drug, or any other condition that may place the patient at risk.
* Patient has a history of other malignancies that have required systemic treatment within the last 2 years or are deemed by the investigator to have a potential to interfere with the safety and efficacy assessment of MRX2843. Patients with treated nonmelanoma skin cancer, in situ carcinoma or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed.
* Patient has received radionuclide treatment within 6 weeks of the first dose of study treatment.
* Patient has received systemic antineoplastic therapy within 14 days of study treatment or 6 weeks for nitrosoureas or mitomycin C. (However, hydroxyurea can be given for the purposes of cytoreduction up to 1 day prior to enrollment, with the exceptions noted above in the inclusion criteria).
* Patient has not fully recovered from acute toxic effects due to all prior therapies, except alopecia and other non-clinically significant AEs prior to enrollment.
* Patient has active clinically significant GvHD.
* Patient has received calcineurin inhibitors within four weeks of study treatment.
* Patient is known to have human immunodeficiency virus infection (HIV).
* Patient has used a small molecular kinase inhibitor or any investigational drug or product within 28 days or 5 half lives, whichever is longer, before study drug dosing.
* Patient has a diagnosis of active hepatitis B or C.
* Patient has an active uncontrolled infection.
* Patient has a history of Type 1 Diabetes (T1D) or is considered at high risk for T1D, where high risk is defined as

  1. Patient has 1 first-degree relative (FDR; defined as parents, offspring or siblings) with T1D AND A1C value > 6.5% or
  2. Patient has 2+FDR with T1D
* Patient has known or suspected history of retinitis pigmentosa or known or suspected familial history of retinitis pigmentosa.
* Patient requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or coumadin-related agents, thrombin or FXa inhibitors, and antiplatelet agents (e.g., clopidogrel). Low dose aspirin (≤ 81 mg/day), low-dose warfarin (≤1 mg/day), and prophylactic Low Molecular Weight Heparin (LMWH) are permitted.
* Patient has congestive heart failure New York Heart Association (NYHA) class 3 or 4, or patient with a history of congestive heart failure NYHA class 3 or 4 in the past, unless a screening echocardiogram performed within 3 months prior to study entry results in a left ventricular ejection fraction that is ≥ 45%.
* Patient has QTcF > 480 ms.
* Patient has had major surgery within 4 weeks of the first dose of study drug.
* The patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects with Dose Limiting Toxicities (DLTs) | Baseline to the end of Cycle 1 (up to 28 days)
Percentage of subjects with Adverse Events (AEs) and Serious Adverse Events (SAEs) graded per National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5 | Baseline up to 14 days after last dose of study treatment (up to approximately 8 months)

SECONDARY OUTCOMES:
Determine Maximum Tolerated Dose (MTD) in mg of MRX-2843 | Baseline to end of Cycle 1 (up to 28 days)
AUC0-t: area under the concentration-time curve from time 0 to the time of the last | Day 1 and Day 23 of Cycle 1 (each cycle is 28 days)
AUC0-inf: area under the concentration-time curve from time 0 to infinity | Day 1 and Day 23 of Cycle 1 (each cycle is 28 days)
AUC0-τ: area under the concentration-time curve from time 0 to tau, where tau is the dosing interval | Day 1 and Day 23 of Cycle 1 (each cycle is 28 days)
Cmax: maximum observed plasma concentration | Day 1 and Day 23 of Cycle 1 (each cycle is 28 days)
Tmax: time to reach maximum observed plasma concentration | Day 1 and Day 23 of Cycle 1 (each cycle is 28 days)
λz: terminal phase elimination rate constant | Day 1 and Day 23 of Cycle 1 (each cycle is 28 days)
t1/2: apparent terminal elimination half-life | Day 1 and Day 23 of Cycle 1 (each cycle is 28 days)
CL/F: apparent total body clearance | Day 1 and Day 23 of Cycle 1 (each cycle is 28 days)
Vz/F: apparent volume of distribution of the terminal phase | Day 1 and Day 23 of Cycle 1 (each cycle is 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda Pauley, MD, Principal Investigator — Emory University, Children's Healthcare of Atlanta; William Blum, MD, Principal Investigator — Emory University; Thomas Alexander, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center, Children's; Joshua Zeidner, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Emory University - WINSHIP Cancer Center, Atlanta, Georgia
  - Emory University, Children's Healthcare of Atlanta, Atlanta, Georgia
  - Memorial Sloan Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No